CLINICAL TRIAL: NCT05544110
Title: Study on the Effect and Mechanism of Individualized and Precise Location Transcranial Magnetic Stimulation Based on Magnetic Resonance Imaging on Post-traumatic Stress Disorder
Brief Title: Precise Transcranial Magnetic Stimulation for Post-traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20222176-F-1
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-02

CONDITIONS: PTSD
Keywords: Transcranial magnetic stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation group (Experimental): Participants receive active transcranial magnetic stimulation.
  Interventions: Device: Active transcranial magnetic stimulation
- Sham stimulation group (Sham Comparator): Participants receive sham transcranial magnetic stimulation.
  Interventions: Device: Sham transcranial magnetic stimulation

INTERVENTIONS:
Device: Active transcranial magnetic stimulation — The coil parallel to the scalp is placed on the target for real and effective stimulation.
  Arms: Active stimulation group
Device: Sham transcranial magnetic stimulation — The coil is placed perpendicular to the scalp above the target for ineffective stimulation.
  Arms: Sham stimulation group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of repetitive transcranial magnetic stimulation under precise localization for post-traumatic stress disorder

DETAILED DESCRIPTION:
Participants who meet the entry conditions and sign the informed consent will be divided into two groups. The stimulation target of each participant will be determined according to MRI. The test group will receive active transcranial magnetic stimulation for 10 consecutive days, and the control group will receive sham stimulation. Symptom severity is assessed by scales and audio and video recordings at baseline, during treatment period and follow-up.Blood samples will also be collected from patients prior to treatment and will be analyzed histologically to explore differences in response to the intervention and biological mechanisms in different subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject, regardless of gender, aged between 18 and 65 years, is admitted to the psychosomatic outpatient department of the First Affiliated Hospital of Air Force Medical University;
* The subject meets the diagnostic criteria of post-traumatic stress disorder in Diagnostic and Statistical Manual of Mental Disorders-5;
* The score of Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 > 33；
* The subject can understand and is willing to strictly abide by the clinical trial protocol and signs the informed consent.

Exclusion Criteria:

* The subject has serious physical diseases or diseases that may affect the central nervous system (such as tumor, syphilis, etc.);
* Patients with PTSD who keep stable on their original medication/psychotherapy for more than 3 weeks before the start of the study or who have not taken the relevant therapeutic medication for more than 2 weeks before the start of the study will be included.Otherwise they will be excluded;
* The subject had previous brain diseases, head trauma, alcoholism, EEG abnormalities, MRI evidence of abnormal brain structure, or family history of epilepsy;
* The subject has contraindications to MRI scanning or transcranial magnetic stimulation treatment, such as metal or electronic instruments (intracranial metal foreign bodies, cochlear implants, cardiac pacemakers, stents and other metal foreign bodies) and space phobia;
* The subject has a history of contact with psychoactive substances or other mental diseases;
* Those at high risk of suicide, or those who have committed suicide or serious self injury and need emergency intervention;
* Pregnant, breastfeeding or planning pregnancy during the trial;
* In the judgment of the investigator, the subject has other conditions that are not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5 scores from baseline to 4 Weeks after the end of the 10 day treatment period | Baseline and Week 4 after the end of the 10 day treatment period
  Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5（PCL-5） is a validated, self-reported instrument assessing PTSD symptom severity over the past week or month period .Possible scores range from 0 to 80 .
  Change = (Week 4 Score -Baseline Score).

SECONDARY OUTCOMES:
Change in Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5 scores scores from baseline to the end of the 10 day treatment period | Baseline and 10 days
  Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5（PCL-5）is a validated, self-reported instrument assessing PTSD symptom severity over the past week or month period .Possible scores range from 0 to 80 .
  Change = (End Score -Baseline Score).
Change in Hamilton Depression Scale scores from baseline to 4 Weeks after the end of 10 day treatment period | Baseline and Week 4 after the end of 10 day treatment period
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
Change in Hamilton Depression Scale（HAMD-17）scores from baseline to the end of 10 day treatment period | Baseline and 10 days
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
Change in Hamilton Anxiety Scale scores from baseline to 4 Weeks after the end of 10 day treatment period | Baseline and Week 4 after the end of 10 day treatment period
  Hamilton Anxiety Scale(HAMA） is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.
Change in Hamilton Anxiety Scale scores from baseline to the end of 10 day treatment period | Baseline and 10 days
  Hamilton Anxiety Scale（HAMA） is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.
Changes of resting state functional connectivity from baseline to the end of the 10 day treatment period | Baseline and 10 days
  Before and after treatment, MRI is performed for each patient to measure the blood oxygen level of each brain region, from which the functional connectivity between brain regions could be statistically obtained, and then the differences of the functional connectivity before and after treatment are compared
Behavioral changes from baseline to the end of the 10 day treatment period | Baseline and 10 days
  PTSD structured interviews will be conducted with participants at baseline and after the treatment. At the same time, audio and video recordings will be made, and data such as expression, language and body movements will extracted for comparison before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huaning Wang, Principal Investigator — Xijing Hospital
Locations (1):
- XIJING Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philip NS, Barredo J, Aiken E, Larson V, Jones RN, Shea MT, Greenberg BD, van 't Wout-Frank M. Theta-Burst Transcranial Magnetic Stimulation for Posttraumatic Stress Disorder. Am J Psychiatry. 2019 Nov 1;176(11):939-948. doi: 10.1176/appi.ajp.2019.18101160. Epub 2019 Jun 24. PMID 31230462
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Koch SB, van Zuiden M, Nawijn L, Frijling JL, Veltman DJ, Olff M. ABERRANT RESTING-STATE BRAIN ACTIVITY IN POSTTRAUMATIC STRESS DISORDER: A META-ANALYSIS AND SYSTEMATIC REVIEW. Depress Anxiety. 2016 Jul;33(7):592-605. doi: 10.1002/da.22478. Epub 2016 Feb 25. PMID 26918313
- [Background] Raij T, Nummenmaa A, Marin MF, Porter D, Furtak S, Setsompop K, Milad MR. Prefrontal Cortex Stimulation Enhances Fear Extinction Memory in Humans. Biol Psychiatry. 2018 Jul 15;84(2):129-137. doi: 10.1016/j.biopsych.2017.10.022. Epub 2017 Nov 6. PMID 29246436
- [Background] Fenster RJ, Lebois LAM, Ressler KJ, Suh J. Brain circuit dysfunction in post-traumatic stress disorder: from mouse to man. Nat Rev Neurosci. 2018 Sep;19(9):535-551. doi: 10.1038/s41583-018-0039-7. PMID 30054570
- [Derived] Zhang Y, Peng Z, Tang N, Zhang Y, Liu N, Lv R, Meng Y, Cai M, Wang H. Efficacy of MRI-guided rTMS for post-traumatic stress disorder by modulating amygdala activity: study protocol for a randomised controlled trial. BMJ Open. 2024 Jul 3;14(7):e081751. doi: 10.1136/bmjopen-2023-081751. PMID 38960463